CLINICAL TRIAL: NCT01044420
Title: mFOLFIRI as the Second Line Chemotherapy for Advanced Esophageal Carcinoma After Failure of 1st Line Treatment of Paclitaxel/DDP : a Phase II Single Center Prospective Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: zhang xiaodong, Peking University, School of Oncology, Department of GI oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLFIRI-AEC2
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-05

CONDITIONS: Advanced Esophageal Carcinoma

ARMS (1):
- mFOLFIRI (Experimental)
  Interventions: Drug: mFOLFIRI

INTERVENTIONS:
Drug: mFOLFIRI — mFOLFIRI irinotecan 130-150mg/m2 iv d1 LV 200 mg/m2 iv 2h d1 5-FU 400 mg/m2 IV d1 5-FU 2.4-3 g/m2 CI 46-h repeat every 2 weeks

SUMMARY:
There are few studies about 2nd line treatment in advanced esophageal carcinoma(AEC), some showed that irinotecan may be effective. The investigators previous study has shown the efficacy and safety of paclitaxel/cisplatin as 1st line treatment, so in this phase II study, the investigators would like to observe the efficacy and safety of Irinotecan/5FU/leucovorin as 2nd line treatment if AEC after failure to 1st treatment of PTX/DDP.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age 18 to 70 years old
* Histologically confirmed esophageal squamous carcinoma,failed to 1st line treatment of paclitaxel/cisplatin
* Unresectable recurrent or metastatic disease
* Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
* Karnofsky performance status ≥70
* Life expectancy of ≥3 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)(within 7 days before enrollment)
* Serum AKP < 2.5 times ULN (within 7 days before enrollment)
* Serum creatinine <1.0 times ULN (within 7 days before enrollment)
* Bilirubin level < 1.0 times ULN (within 7 days before enrollment)
* WBC>4,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl(within 7 days before enrollment)
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever>38℃；
* Good compliance

Exclusion Criteria:

* More than 1 Previous systemic therapy for metastatic esophageal squamous carcinoma
* Known hypersensitivity to irinotecan
* Only with Brain or bone metastasis
* Tumor with length≥10cm, liver metastasis covers more than 50% of liver,or lung metastasis covers more than 25% of lung
* No measurable lesions, eg. pleural fluid and ascites
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry
* Heart failure or other sever organ dysfunction, eg. coronary artery disease, myocardial infarction within the last 6 months or
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Chronic diarrhea
* Mentally abnormal or disable cognition,including CNS metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 year
adverse events | after each cycle of chemotherapy

SECONDARY OUTCOMES:
progression-free survival | 1year
response rate | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: shen lin, MD, Study Chair — peking university, school of oncology, department of GI oncology; zhang xiaodong, MD, Principal Investigator — Peking University, school of oncology, department of GI oncology
Locations (1):
- Zhang Xiaodong, Beijing, Beijing Municipality, China